CLINICAL TRIAL: NCT00013845
Title: Evaluation and Treatment of Patients With Epilepsy
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010139; 01-N-0139
Record Dates: First submitted 2001-03-30; First posted 2001-04-02 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-06-26

CONDITIONS: Epilepsy
Keywords: Seizures; Anti-Epileptic Drugs; Pharmacotherapy; Neuropsychology; Temporal Lobe Epilepsy; Frontal Lobe Epilepsy; Complex Partial Seizures; Grand Mal Seizures; Generalized Seizures; Epilepsy
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsy, Temporal Lobe; Epilepsy, Frontal Lobe; Epilepsy, Tonic-Clonic

SUMMARY:
This protocol has three purposes: 1) to screen patients with seizures for participation in research studies of NINDS s Clinical Epilepsy Section (CES), 2) to follow the natural course of seizure disorders, and 3) to train CES fellows in evaluating and treating epilepsy. Only standard diagnostic tests and treatments will be used in this study.

Patients of any age with seizures who are referred to CES may participate in this study. At the end of the study, patients may be discharged to the care of their referring physician, offered participation in another NINDS research protocol, or followed for teaching purposes.

Participants will undergo standard diagnostic procedures used to determine the type of their seizures, what part of the brain they are coming from, what is causing them, and whether standard drug treatments can help them. These may include some or all of the following:

* Physical and neurological examination
* Neuropsychological tests tests of learning and memory
* Electroencephalography (EEG) brain wave recording
* Evoked potentials tests of nerve reactions to lights and sounds
* Polysomnography simultaneous recordings of brain waves, breathing and eye movements
* Video-EEG monitoring simultaneous recording of seizures using a video camera and brain waves
* Video-EEG monitoring with extra electrodes to record muscle activity, breathing and eye movements for analyzing sleep patterns
* Imaging studies, such as magnetic resonance imaging (MRI) and positron emission tomography (PET) scans to examine the structure and function of the brain
* Frequent blood tests to measure blood levels of anti-seizure drugs

DETAILED DESCRIPTION:
Objectives: To evaluate patients with epilepsy

Study Population: adults and children with epilepsy

Design: In this protocol we will use standard clinical studies, including neurologic examination, antiepileptic drug levels, clinical neurophysiology (EEG, EMG, evoked potentials, simultaneous Video-EEG monitoring, polysomnography), computed tomography, structural functional, and spectroscopic magnetic resonance imaging, and other studies, such as FDG-PET (performed by nuclear medicine as a clinical procedure) and neuropsychological testing, to evaluate patients referred for uncontrolled or suspected seizures. Tests will be performed in patients when clinically indicated. The protocol will be used to screen patients for inclusion in other protocols, follow the natural history of seizure disorders, and train fellows in the evaluation and treatment of epilepsy. Both inpatients and outpatients will be studied. Standard clinical evaluation and drug treatment of epilepsy is performed under this protocol.

Outcome Measures: clinical characteristics of epilepsy

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients older than 2 years referred to the Clinical Epilepsy Section will be included. DPA assignment for adults without consent capacity is required at the time of enrollment.

EXCLUSION CRITERIA:

None.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1278 (Actual)
Dates: Start 2001-05-01; Study Completion 2018-06-26

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Inati, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baker GA, Nashef L, van Hout BA. Current issues in the management of epilepsy: the impact of frequent seizures on cost of illness, quality of life, and mortality. Epilepsia. 1997;38 Suppl 1:S1-8. doi: 10.1111/j.1528-1157.1997.tb04511.x. PMID 9092951
- [Background] Begley CE, Famulari M, Annegers JF, Lairson DR, Reynolds TF, Coan S, Dubinsky S, Newmark ME, Leibson C, So EL, Rocca WA. The cost of epilepsy in the United States: an estimate from population-based clinical and survey data. Epilepsia. 2000 Mar;41(3):342-51. doi: 10.1111/j.1528-1157.2000.tb00166.x. PMID 10714408
- [Background] Hanai T. Quality of life in children with epilepsy. Epilepsia. 1996;37 Suppl 3:28-32. doi: 10.1111/j.1528-1157.1996.tb01816.x. PMID 8681908